CLINICAL TRIAL: NCT01341834
Title: A Safety and Tolerability Study of RAD001 (mTOR Inhibitor) in Combination With Two Dosing Schedules of LBH589B (Histone Deacetylase Inhibitor) in Solid Tumors/ Lymphomas With Enrichment for EBV-Driven Tumors
Brief Title: Safety and Tolerability Study of RAD001 and LBH589 in All Solid Tumors With Enrichment for EBV Driven Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-01-ST_ECRU
Record Dates: First submitted 2011-04-21; First posted 2011-04-26 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Nasopharyngeal Carcinoma, Lymphomas, Any EBV+ Solid Tumour
Keywords: Nasopharyngeal carcinoma, antiangiogenesis, HDACi, mTOR, Phase Ib
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Lymphoma; Hereditary Sensory and Autonomic Neuropathies | interventions — Panobinostat; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LBH589-RAD001 (Experimental): LBH589-RAD001, single arm dose finding study
  Interventions: Drug: LBH589 and RAD001

INTERVENTIONS:
Drug: LBH589 and RAD001 — Dose escalation of LBH589 tablets (5 and 10 mg) and RAD001 tablets (2.5, 5 mg and 10mg)

SUMMARY:
The purpose of this study is:

1. To determine the optimal recommended phase II dose of two investigational study drugs, LBH589 and RAD001, given in combination in all solid tumors (With enrichment for EBV-Driven tumors).
2. To determine the pharmacokinetic profile of RAD001 in combination with two schedules of LBH589.
3. To assess the preliminary anti-tumor activity of RAD001 and LBH589.

This study will also be exploring the hypothesis that HDACi and mTOR inhibitors abrogate the effects of key viral proteins, and switch the virus from a latent proliferative phase to a lytic phase. Immunologic correlates will also be examined to ascertain T-cell subpopulations and expression of HLA class molecules. DCE-MRI will be subsequently employed in dose expansion to examine antiangiogenic effects.

DETAILED DESCRIPTION:
Dose escalation phase 1B of the study will evaluate the safety and tolerability of RAD001 in combination with LBH589 in all solid tumors, lymphomas; and enriched for EBV driven tumors. The phase 2 component will be a single arm, non-randomized study restricted to nasopharyngeal carinoma only (endemic type).

A "3+3" dose escalation design will be adopted. Patients will start taking LBH589 three times a week and will have a run in period of one week, followed by continous administration of RAD001 from week 2. Pharmacokinetic assessments will be done on day 1 of LBH589 administration and day 1 of concurrent administration of LBH589 + RAD001. ON day 31, there will be a one week drug holiday. This is done to explore the eliminaition kinetics from steady state,as well as the durability of target modulation.

AEs of patients will be monitored closely. In the event of grade 3/4 toxicity, the cohort will be expanded to 6. Dose escalation of LBH589/RAD001 may proceed until the maximum tolerated dose (MTD)is reached. Once the MTD is established, an expasion cohort comprising 20 EBV driven tumors will open at two different LBH589 dose schedules.

Treatment will be continued until progression of disease, unacceptable toxcity, or discontinuation criterion is met.

ELIGIBILITY:
Inclusion criteria

1. Patients with histologically or cytologically confirmed solid malignancy or lymphoma that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective.

   For enrichment and dose expansion phase only:

   Only patients with EBV-related tumors, including all nasopharyngeal carcinoma, as well as tumors known to be EBV-related which include (but are not limited to) gastric carcinoma (10-15%), lymphoma. These tumors (NPC excluded) should have:

   i)EBER in situ hybridisation on paraffin samples/ circulating tumor cells; or ii)Elevated pre-treatment serum EBV viral titres
2. Patients who have had prior treatment with mTOR inhibitors and HDAC inhibitors will be allowed ONLY in the dose escalation phase
3. Age ≥ 21 years old.
4. Performance status of ≤ 2 (ECOG scale).
5. Target lesion on spiral CT or MRI scan must have at least one diameter > 1 cm (on conventional CT scan the indicator lesion must have at least one diameter > 2 cm) (for dose expansion).
6. Adequate bone marrow reserve: absolute granulocyte count > 1 x 109/L, hemoglobin > 8 g/dL and platelet count >100,000/dL.
7. Adequate hepatic function (serum total bilirubin level < 1.5 x ULN; alanine transaminase (ALT) and aspartate transaminase (AST) less than 3 times ULN.
8. Adequate renal function (creatinine < 1.5 times ULN).
9. Normal ECG at baseline - with no significant conduction abnormalities and a QTc ≤ 450.
10. Left Ventricular Ejection Fraction ≥ 50% as assessed by MUGA scan or echocardiography at screening.
11. No concurrent use of investigational antineoplastic therapy.
12. No medical problems severe enough to prevent compliance with the study requirements
13. Negative pregnancy test (urinary β-HCG) at screening (applicable to women of child bearing potential who are sexually active).
14. Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Known brain metastases (locally advanced NPC with direct extension to central nervous system is permissible).
2. Chemotherapy (in the case of nitrosoureas and mitomycin C within 6 weeks), radiotherapy, immunotherapy within 4 weeks before study drug administration.
3. Patients receiving chronic immunosuppressive treatment with high dose corticosteroids (tailing doses or low doses are acceptable) or another immunosuppressive agent;
4. Patients with uncontrolled diabetes (fasting glucose > 2x ULN);
5. History of uncontrolled heart disease (unstable angina, congestive heart failure, myocardial infarction within preceding 12 months, clinically significant rhythm or conduction abnormality such as second and third degree heart block, congenital long QT syndrome, obligate use of a cardiac pacemaker. Patients with QTc at screening > 450 ms.
6. Subjects taking medications known to have a risk of causing causing QTc prolongation and Torsades de Pointes (risk group 1 as indicated on webpage: http://www.torsades.org).
7. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat treatment.
8. Patients with impairment of GI function or GI disease that may significantly alter panobinostat absorption.
9. Patients with unresolved diarrhea of grade 2 and above.
10. Patients with a known history of Hepatitis B, C and HIV seropositivity.
11. Patients with an active bleeding diathesis;
12. Subjects with Grade ≥ 2 neuropathy at baseline.
13. For patients undergoing magnetic resonance imaging (MRI) studies (including DCE-MRI, BOLD-MRI and DWI-MRI) in the expansion cohort:

    1. Contraindications to MRI, e.g. contraindicated metal implants
    2. Patients with poor antecubital fossa venous access.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Weekly evaluation for the first 5 weeks (DLT period), and continued follow up until patients come off trial due to toxicity or progressive disease
  Patients will be followed closely for toxicities in the first cycle where they would have weekly consultations visit. After the first cycle, consultation visits will be once every 2 weeks or once a month depending on how well the patient is tolerating the treatment.
  The following safety assesments will be done on every visit; Vital signs and physical examination Haematology and blood chemistry Cardiac monitoring EBV DNA titre (for patients with EBV Driven tumors recording of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Tumor response | Every 2 months until disease progression or withdrawal from study - average of 6 - 12 months
  Tumor response will be evaluated at the end of every 8-weeks of treatment. Treatment will continue until one of the following occur; disease progression, unacceptable toxicity, death, or withdrawal from study. Best response (according to RECIST), as well as progression free survival will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tan Shao Weng, Principal Investigator — National Cancer Center Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore